CLINICAL TRIAL: NCT03376022
Title: Attitudes and Knowledge of Oral Health Among Nursing Personnel
Status: Completed | Type: Observational
Sponsor: Dalarna County Council, Sweden (Other)
Responsible Party: Principal Investigator, Kristina Edman, Principal investigator, Dalarna County Council, Sweden
Other Study IDs: Nursing personnel, oral health
Record Dates: First submitted 2017-10-20; First posted 2017-12-18 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Knowledge, Attitudes, Practice; Attitude; Oral Health
Keywords: Attitudes; Knowledge; Oral Health; Nursing personnel
MeSH Terms: conditions — Behavior | interventions — Health Knowledge, Attitudes, Practice

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Attitudes, knowledge — To investigate attitudes and knowledge to oral Health and oral care

SUMMARY:
Oral Health care has been shown to have low priority among nursing personnel, especially among personnel with shorter education.

DETAILED DESCRIPTION:
As the population gets older and keep their natural teeth high up in age, in most cases throughout life, it is of importance to help the older maintain a good oral health when the cognitive functions and physical ability decreases. In 1999, a new dental care system was introduced with the aim to offer elderly with long-term need for extensive care, home visits for oral health assessment and, if necessary, be offered the necessary dental care. The aim was also to offer nursing personnel education and training in dental health and oral care, in order to provide and perform oral care. The effect of the education program has never been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Nursing personnel in nursing home for elderly
* Must be able to read and understand Swedish

Exclusion Criteria:

- None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All nursing personnel in nursing home for elderly in the County of Dalarna Sweden.
Sampling Method: Probability Sample
Enrollment: 4500 (Actual)
Dates: Start 2018-05-22 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Attitudes to Oral Health and oral care | February 2019
  A questionnaire, Dental Coping Beliefs Scale (DCBS) will be used to investigate attitudes to, and knowledge of oral health among nursing staff caring for home-dwelling older people. DCBS investigates three dimensions; Locus of control (internal and external), self-efficacy and oral-health care believes.
  Apart from descriptive statistics, a logistic regression model will be used to analyze the relationship between the sum scores for the factors Oral health care beliefs, Internal locus of control, External locus of control and background variables (age, work experience and earlier adjunct education).

CONTACTS AND LOCATIONS:
Overall Officials: Kristina A Edman, PhD, Principal Investigator — Dalarna Public Dental Health
Locations (1):
- Kristina Edman, Falun, Dalarna County, Sweden

IPD SHARING:
Plan to Share IPD: No